CLINICAL TRIAL: NCT06466239
Title: Acute Effect of Self-PNF Stretching on Chest Mobility, Posterior Muscle Chain Mobility and Respiratory Functions in Caregivers of Children With Developmental Delays
Brief Title: PNF Method for Those Working in Special Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Collaborators: Istanbul Gedik University (Other)
Responsible Party: Principal Investigator, ebrar atak, Asst. Prof., Medipol University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: PNFEffectsForCaregiver
Record Dates: First submitted 2024-06-07; First posted 2024-06-20 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Caregiver Burden
Keywords: maintenance burden; PNF technique; rehabilitation worker
MeSH Terms: conditions — Caregiver Burden | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PNF Stretching Group (Experimental): The PNF stretching method for each muscle was applied to the athlete in the form of self-stretching by the participant, with the direct treatment concept of hold and relax technique, with the training of a specialist physiotherapist. The muscle to be stretched (the antagonist muscle for the pattern - the muscle that causes the limitation) was first brought to the position where it could be extended, and at that point, the stretched muscle was contracted submaximally (65% of the intensity determined according to the Stretch Intensity Scale) for 5 seconds, causing isometric contraction. Then, the athlete was given 5 relax commands for the tense muscle. Then, the stretched muscle was stretched as far as it could go, and the muscle that needed to be stretched was passively stretched for 20 seconds (1 set). After a 5-second rest interval, the method was repeated and 8 sets (lasting 4 minutes) were performed for 1 muscle. Stretching was done on the hamstring muscle.
  Interventions: Other: PNF Stretching
- Static Stretching Group (Other): Classical static stretching was applied to the hamstring muscle in the same position for 30 seconds each, 8 repetitions, a total of 4 minutes for one leg and 8 minutes for both legs, in the stance position of PNF stretching.
  Interventions: Other: Static Stretching

INTERVENTIONS:
Other: PNF Stretching — PNF was applied to the hamstring muscle, with a 1-day washout period in between.
  Arms: PNF Stretching Group
Other: Static Stretching — Static stretching was applied to the hamstring muscle, with a 1-day washout period in between.
  Arms: Static Stretching Group

SUMMARY:
The aim of the study was to examine the acute effect of self-proprioceptive neuromuscular facilitation (PNF) stretching on chest mobility, posterior muscle chain mobility and respiratory functions in caregivers of children with developmental delays. In the study: 1. Does self-PNF stretching have an effect on chest mobility and posterior muscle chain mobility in caregivers of children with developmental delay? 2. Does self-PNF stretching have an effect on respiratory functions in caregivers of children with developmental delays? The questions were answered.

DETAILED DESCRIPTION:
A cross-over randomized controlled study was designed with 30 caregivers of children with developmental disabilities. Using the online randomization method, caregivers were first assigned to either the PNF stretching group or the static stretching group. Before and after the application, rib cage mobility was evaluated by chest circumference measurement, hamstring muscle mobility by popliteal angle measurement, lumbar region mobility by Schober Test, posterior muscle chain mobility by Finger-Floor Distance Measurement Test, and respiratory functions by Respiratory Function Test. The caregiver, who entered a 1-day cleansing period, repeated the evaluation and technique application with the stretching technique that was not applied the next day.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study
* No history of infection or flare in the previous 4 weeks
* Participants who have not been included in another clinical trial in the last month
* Those whose knee flexion angle is 15 degrees and above in the hamstring muscle shortness test

Exclusion Criteria:

* Vestibular disorders, participants with known balance impairment within the past three months due to concussion
* Those with musculoskeletal system problems in their lower extremities
* Those who had lower extremity and thorax surgery in the last year
* Those with metabolic diseases

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-11-04 (Actual); Primary Completion 2024-03-12 (Actual); Study Completion 2024-06-06 (Actual)

PRIMARY OUTCOMES:
Chest Mobility Measurement 1- Axillary region | Duration of change in 1 day.
  Normal resting tidal volume, chest width during maximum inspiration and maximum expiration were measured from the axillary region with a tape measure and recorded in centimeters.
Chest Mobility Measurement 2- Xiphoid region | Duration of change in 1 day.
  Normal resting tidal volume, chest width during maximum inspiration and maximum expiration were measured from the xiphoid (epigastric) region with a tape measure and recorded in centimeters.
Chest Mobility Measurement 3- Subcostal region | Duration of change in 1 day.
  Normal resting tidal volume, chest width during maximum inspiration and maximum expiration were measured from the subcostal region with a tape measure and recorded in centimeters.

SECONDARY OUTCOMES:
Popliteal Angle Measurement | Duration of change in 1 day.
  Hamstring muscle flexibility measurement. A digital goniometer was used.
Schober Test | Duration of change in 1 day.
  Lumbar mobility was evaluated with the Schober Test. A tape measure was used in the testing procedure.
Posterior muscle chain mobility measurement | Duration of change in 1 day.
  Posterior muscle chain mobility was evaluated with the Finger-Floor Distance Test. A tape measure was used in the testing procedure.
FVC Measurement | Duration of change in 1 day.
  Respiratory Function Test. The COSMED microQuark spirometer used. Lung volume was evaluated.
FEV1 Measurement | Duration of change in 1 day.
  Respiratory Function Test. The COSMED microQuark spirometer used. Lung volume was evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Ebrar Atak, Yalova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
It will be evaluated if the researchers are contacted via their e-mail addresses.

REFERENCES:
- [Background] Reiner M, Tilp M, Guilhem G, Morales-Artacho A, Nakamura M, Konrad A. Effects of a Single Proprioceptive Neuromuscular Facilitation Stretching Exercise With and Without Post-stretching Activation on the Muscle Function and Mechanical Properties of the Plantar Flexor Muscles. Front Physiol. 2021 Sep 14;12:732654. doi: 10.3389/fphys.2021.732654. eCollection 2021. PMID 34594241